CLINICAL TRIAL: NCT00855023
Title: Tibiofemoral Alignment: Contributing Factors to Noncontact Anterior Cruciate Ligament Injury
Brief Title: Knee Alignment Contributions to Anterior Cruciate Ligament (ACL) Injury
Status: Completed | Type: Observational
Sponsor: The Orthopaedic Center, Maryland (Other)
Responsible Party: Principal Investigator, Barry P. Boden, MD, M.D., researcher, The Orthopaedic Center, Maryland
Other Study IDs: 07-08-229-147
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2009-03

CONDITIONS: Knee Injuries
Keywords: anterior cruciate ligament; Knee Joint
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asymptomatic Volunteers: healthy volunteer athletes and excluded those who had any of the following criteria: 1) counter-indications to magnetic resonance imaging (e.g., pregnancy or postsurgical hardware [plates, screws, aneurysm clip, implanted cardiac pacemaker, etc.]); (2) relevant medical problems (e.g., connective tissue problems, paralyzed hemidiaphragm, morbid obesity, claustrophobia, etc.); (3) clinical signs of an impairment or abnormality in the knee (e.g., abnormal range of motion, muscle weakness, or malalignment); (4) injury to the knee that required medical attention; (5) previous surgery on the knee; or (6) current pain in the knee.

SUMMARY:
This study evaluates the the anatomic factors of the knee that may predispose to ACL injury.

DETAILED DESCRIPTION:
Despite intense study of anterior cruciate ligament injury during the past three decades, the mechanisms of this injury have not been clearly defined. A recent study by the Principle Investigator identified differences in leg alignment when a single leg landing during a sports activity resulted in a torn ACL and when it did not (provocative versus control alignment, respectively).

The purpose of the study is to quantify the tibiofemoral alignment in the lateral compartment of the knee in the provocative landing position and the control landing position. in order to elucidate possible mechanisms of ACL injury Material and Methods: 25 normal controls will be recruited from the greater Washington DC population. Magnetic resonance images in the sagittal plane will be acquired for a single leg of each subject. These images will cover the lateral compartment of the knee and will be acquired with the leg in three positions, one that emulates the injury position, one that exagerrates the injury position, and one that emulates the control landing position. Statistical analysis of the measurements between the provocative, exagerrated provocative, and control positions will then be performed.

These insights could then be applied to improving training focused on reducing the incidences of ACL rupture; improving bracing designs to help athletes most at risk of ACL rupture or those recovering from ACL injury/surgery; and improving ACL replacement surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls
* Ages 18-45 years old

Exclusion Criteria:

* Previous knee injury or surgery
* Metal implants in body

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteer athletes and excluded those who had any of the following criteria: 1) counter-indications to magnetic resonance imaging (e.g., pregnancy or postsurgical hardware [plates, screws, aneurysm clip, implanted cardiac pacemaker, etc.]); (2) relevant medical problems (e.g., connective tissue problems, paralyzed hemidiaphragm, morbid obesity, claustrophobia, etc.); (3) clinical signs of an impairment or abnormality in the knee (e.g., abnormal range of motion, muscle weakness, or malalignment); (4) injury to the knee that required medical attention; (5) previous surgery on the knee; or (6) current pain in the knee.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Measurement of anatomy of knee | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Barry P Boden, MD, Principal Investigator — The Orthopedic Center
Locations (1):
- Open MRI of Washington, Rockville, Maryland, United States

REFERENCES:
- [Background] Boden BP, Torg JS, Knowles SB, Hewett TE. Video analysis of anterior cruciate ligament injury: abnormalities in hip and ankle kinematics. Am J Sports Med. 2009 Feb;37(2):252-9. doi: 10.1177/0363546508328107. PMID 19182110
- [Derived] Boden BP, Breit I, Sheehan FT. Tibiofemoral alignment: contributing factors to noncontact anterior cruciate ligament injury. J Bone Joint Surg Am. 2009 Oct;91(10):2381-9. doi: 10.2106/JBJS.H.01721. PMID 19797573